CLINICAL TRIAL: NCT06666556
Title: Bowel Preparation in Colonoscopy: Lactulose Vs Polyethyleneglycol, Randomized Double-blind Comparative Clinical Trial, Multicenter Study.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Roberto Ulises Cruz Neri, M. C. Roberto Cruz Neri (Master in cience, medical staff Coloproctology Department Hospital Civil Fray Antonio Alcalde), Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 151/24
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer Screening
Keywords: colorectal; colorectal cancer; colorectal cancer screening; colonoscopy; polyethylenglycol; lactulose
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Lactulose; alginate-polyethylene glycol acrylate

STUDY DESIGN:
Intervention Model Description: multicenter single-blind randomized clinical trial study
Who Masked: Care Provider
Masking Description: The main investigators will be in charge of randomizing all the patients ellegible for this protocol, and the care providers and endoscopists will be masked when it comes to knowing to which arm of the study each patient belongs to, untill the moment they need to perform the colonoscopy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Bowel preparation with lactulose before de colonoscopy (Active Comparator): Patients will be randomized and assigned the bowel preparation the day that provide them the day of the colonoscopy
  Interventions: Combination Product: Bowel preparation before colonoscopy
- Bowel preparation with plyethylenglycol before the colonoscopy (Active Comparator): Patients will be randomized and assigned the bowel preparation the day that provide them the day of the colonoscopy
  Interventions: Combination Product: Bowel preparation before colonoscopy

INTERVENTIONS:
Combination Product: Bowel preparation before colonoscopy — In this multicenter single-blind randomized clinical trial study we will provide each patient that meets our inclusion criteria a randomized folio to include them in one of both arms in our protocol, meaning one of the groups and the bowel preparation assigned to perform the colonoscopy, they will be explained the benefits and minimum risks of participating and they will also be asked to sign an informed consent form so we can continue with the colonoscopy and collect all the data we need for our protocol and the analysis of the variables.
  Other Names: Lactulose
  Arms: Bowel preparation with lactulose before de colonoscopy
Combination Product: Bowel preparation before colonoscopy — In this multicenter single-blind randomized clinical trial study we will provide each patient that meets our inclusion criteria a randomized folio to include them in one of both arms in our protocol, meaning one of the groups and the bowel preparation assigned to perform the colonoscopy, they will be explained the benefits and minimum risks of participating and they will also be asked to sign an informed consent form so we can continue with the colonoscopy and collect all the data we need for our protocol and the analysis of the variables.
  Other Names: Polyethylenglycol
  Arms: Bowel preparation with plyethylenglycol before the colonoscopy

SUMMARY:
The goal of this clinical trial it is to bowel the instestinal preparation with lactulose vs poliethylenglicol as better agent to have a quality colonoscopy and demostrate that lactulose is most efective, has a good tolerance and the patient would have a better satisfaction, so the question is:

wich is the eficancy of lactulose in comparision with thepoliethylenglycol in the intestinal preparation for the colonoscopy?

DETAILED DESCRIPTION:
A bowel preparation is fundamental before making a colonoscopy, letting us realize a correct exploration in all the bowel. The main method of cleaning would be fast, safe and getting a high grade of visualizing to do a quality colonoscopy.

Actually there are a lot of methods or products of cleaning the bowel. A good cleaning have a lot of successful choosing a good product to do it and having a good diet before the colonoscopy.

There are a lot of scales about the cleaning in the colonoscopy, having a good bowel preparation increase the capacity of the detection of polyps, decrease the time of the colonoscopy and getting better the cost and efficiency.

The colonoscopy plays a crucial role in the screening and treatment of colorectal cancer. It is an optimal procedure to identify precancerous lesions. polyps and recommended for screening people with risk factors, such as a family history of polyps or cancer.

Bowel preparation is a crucial aspect in colonoscopy due to its direct relationship with the quality of the procedure. Many patients find bowel preparation to be the most uncomfortable part of the examination, so ensuring that it is safe, extremely efficient, reliable, convenient and tolerable enough to ensure that patients will not be able to complete it or wish to undergo future procedures, associating this with the bad taste of the agents used and the adverse events produced.

Ignorance of the importance of adequate bowel preparation and cleansing explains poor adherence to instructions, and increases the rate of inadequate bowel preparation.

The health team must provide correct and clear information that improves patient adherence. The importance of compliance with the indications and the impact of adequate intestinal cleansing on the findings and results of colonoscopy should be emphasized.

The cleaning systems used in colonoscopy must allow more than 90% of the mucosal surface to be explored. Furthermore, the drugs used must be well tolerated by the patient and not cause side effects. Therefore, the ideal colonoscopy preparation should combine efficacy, excellent tolerance, and minimal adverse effects.

The use of oral bowel preparations may induce strong peristalsis, cramps, bloating, diarrhea and other symptoms. Intolerance to the preparation is common and is usually associated with the volume of liquid consumed and the taste of the solution.

Polyethyleneglycol (Muvinlax(r) or Nulytely is a non-absorbable electrolyte solution and does not induce electrolyte mucus secretion or significantly reduce fluid exchange in the colonic lumen. It has been shown to be non-toxic and can be ingested in large quantities without dangerous effects. Its use is relatively safe in patients with kidney failure, cirrhosis or congestive heart failure.

Bowel preparation with polyethyleneglycol represents the most used formula in our environment. Among the recognized limitations associated with its application are: the large amount of volume to be ingested (4 L), which makes it impossible to administer it to elderly people with swallowing difficulties, it is also poorly tolerated by patients and has been associated with medical complications, among which can be mentioned: vomiting, abdominal distension, abdominal pain, nausea, Mallory Weiss syndrome, esophageal perforation, bronchoaspiration, toxic colitis, pancreatitis induced by polyethyleneglycol.

Lactulose (Duphalac (r)) is a disaccharide, semi-synthetic derivative of lactulose. It is absorbed and undergoes bacterial action, which causes fermentation, acidifying the environment and causing acceleration of intestinal transit, stimulating motility. Another consequence of acidification is the increase in osmotic pressure within the lumen of the colon, proportional to the dose. Regarding the dose, 120 ml are diluted with juice or clear water until completing 1000 ml, swallowing the entire volume in 1 hour The preparation regimen has a significant impact on the quality of intestinal cleansing. Traditionally, preparation is done one day before a colonoscopy.

ELIGIBILITY:
* Inclusion Criteria:
* Patients with indication for colonoscopy in our coloproctology service
* Both women and men
* Patients within an age range of 18-79 years
* Patients who agree having a colonoscopy and who sign the informed consent to participate in the protocol

Exclusion Criteria:

* Patients under 18 or over 80 years old
* All patients that won´t like to participate in the protocol or won´t sign the informed consent
* Pregnant women
* Patients with a medical record of colonic resection, ostomy status, severe cardiopulmonary and renal diseases, major psychiatric disorders, therapeutic colonoscopy or any contraindications for colonoscopy
* Non compliance with the colonic preparation regimen
* Active bleeding during the procedure
* Patients with a known diagnosis of colorectal cancer

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Score of the bowel cleaness | From date of randomization until the colonoscopy is done, assessed up to July 2025.
  It would be evaluated using a standardized scoring system, such as the BBPS scale.

SECONDARY OUTCOMES:
Tolerability | From date of randomization until the colonoscopy is done, assessed up to July 2025.
  Adverse symptoms and general tolerance of patients towards each bowel preparation will be recorded.
Gastrointestinal side effects | From date of randomization until the colonoscopy is done, assessed up to July 2025.
  Any gastrointestinal side effects experienced by patients during the bowel preparation process will be recorded.
Patient Satisfaction and Palatability | From date of randomization until the colonoscopy is done, assessed up to July 2025.
  Data will be collected on overall patient satisfaction and palatability of the agent with the bowel preparation process using a subjective rating scale.

CONTACTS AND LOCATIONS:
Locations (3):
- Mexico (3):
  - Antigüo Hospital Civil de Guadalajara "Fray Antonio Alcalde", Guadalajara, Jalisco
  - Nuevo Hospital Civil de Guadalajara "Juan I. Menchaca", Guadalajara, Jalisco
  - IMSS Hospital General Regional 220 "José Vicente Villada", México, Toluca de Lerdo

REFERENCES:
- [Background] Varea-Calderón V, Martín de Carpi J. Videocolonoscopia: técnica e indicaciones. An Pediatría Contin. el 1 de febrero de 2008;6(1):42-4.
- [Background] Herraiz M. [Colonoscopy with carbon dioxide insufflation: luxury or neccesity?]. Gastroenterol Hepatol. 2013 Jan;36(1):43-7. doi: 10.1016/j.gastrohep.2012.06.002. Epub 2012 Dec 4. Spanish. PMID 23218772
- [Background] Reumkens A, Rondagh EJ, Bakker CM, Winkens B, Masclee AA, Sanduleanu S. Post-Colonoscopy Complications: A Systematic Review, Time Trends, and Meta-Analysis of Population-Based Studies. Am J Gastroenterol. 2016 Aug;111(8):1092-101. doi: 10.1038/ajg.2016.234. Epub 2016 Jun 14. PMID 27296945
- [Background] Pan H, Zheng XL, Fang CY, Liu LZ, Chen JS, Wang C, Chen YD, Huang JM, Zhou YS, He LP. Same-day single-dose vs large-volume split-dose regimens of polyethylene glycol for bowel preparation: A systematic review and meta-analysis. World J Clin Cases. 2022 Aug 6;10(22):7844-7858. doi: 10.12998/wjcc.v10.i22.7844. PMID 36158495
- [Background] Martel M, Barkun AN, Menard C, Restellini S, Kherad O, Vanasse A. Split-Dose Preparations Are Superior to Day-Before Bowel Cleansing Regimens: A Meta-analysis. Gastroenterology. 2015 Jul;149(1):79-88. doi: 10.1053/j.gastro.2015.04.004. Epub 2015 Apr 8. PMID 25863216
- [Background] Arenas M, Pérez-Arellano E. Colonoscopy preparations: electrolyte imbalances and precautions in the fragile patients. Rev Andal Patol Dig. el 30 de abril de 2024;47(2):66-71.
- [Background] Lezama-de-Luna JF, Manrique MA, Chávez-García MÁ, Pérez-Corona T, Gómez-Peña-Alfaro NS, Pérez-Valle E, et al. Evaluación de la eficacia y tolerabilidad de tres esquemas de preparación de colon.
- [Background] Gaballa S, Naguib Y, Mady F, Khaled K. Polyethylene glycol: Properties, applications, and challenges. J Adv Biomed Pharm Sci. el 21 de diciembre de 2023;0(0):26-36
- [Background] Murcio-Pérez E, Téllez-Ávila. F. Opciones de preparación para colonoscopia. Endoscopia. el 1 de enero de 2011;24(1):23-31.
- [Background] Ia I, Ma Á. Preparación intestinal para la colonoscopia en pacientes con diferentes patologías.
- [Background] Quintero E, Alarcon-Fernandez O, Jover R. [Colonoscopy quality control as a requirement of colorectal cancer screening]. Gastroenterol Hepatol. 2013 Nov;36(9):597-605. doi: 10.1016/j.gastrohep.2013.02.005. Epub 2013 Jun 12. Spanish. PMID 23769425
- [Background] Menacho AM, Reimann A, Hirata LM, Ganzerella C, Ivano FH, Sugisawa R. Double-blind prospective randomized study comparing polyethylene glycol to lactulose for bowel preparation in colonoscopy. Arq Bras Cir Dig. 2014 Jan-Mar;27(1):9-12. doi: 10.1590/s0102-67202014000100003. PMID 24676290
- [Background] Sánchez-del-Río A, Pérez-Romero S, López-Picazo J, Alberca-de-las-Parras F, Júdez J, León-Molina J, et al. Indicadores de calidad en colonoscopia. Procedimiento de la colonoscopia. Rev Esp Enfermedades Dig. 2018;110(5):316-26.
- [Background] Hammami A, Elloumi H, Bouali R, Elloumi H. Clinical practice standards for colonoscopy. Tunis Med. 2021 Octobre;99(10):952-960. PMID 35288895
- [Background] Cerna-Cardona J, Peláez-Luna MC, Casillas-Guzmán GB, Sánchez-Chávez X, Casanova-Lara AI, Espino-Cortés H, et al. Guía de endoscopia en enfermedad inflamatoria intestinal. Endoscopia. marzo de 2021;33(1):22-44.
- [Background] Yamamoto-Furusho JK, Bosques-Padilla F, de-Paula J, Galiano MT, Ibanez P, Juliao F, Kotze PG, Rocha JL, Steinwurz F, Veitia G, Zaltman C. Diagnosis and treatment of inflammatory bowel disease: First Latin American Consensus of the Pan American Crohn's and Colitis Organisation. Rev Gastroenterol Mex. 2017 Jan-Mar;82(1):46-84. doi: 10.1016/j.rgmx.2016.07.003. Epub 2016 Dec 13. English, Spanish. PMID 27979414
- [Background] Kim SY, Kim HS, Park HJ. Adverse events related to colonoscopy: Global trends and future challenges. World J Gastroenterol. 2019 Jan 14;25(2):190-204. doi: 10.3748/wjg.v25.i2.190. PMID 30670909
- [Background] Ramírez-Quesada W, Vargas-Madrigal J, Alfaro-Murillo O, Umaña-Solís E, Campos-Goussen C, Alvarado-Salazar M, et al. Indicadores de calidad para la realización de colonoscopia. Acta Médica Costarric. marzo de 2019;61(1):37-42.
- [Background] Church J. Colonoscopy: what are we missing? Surg Oncol Clin N Am. 2014 Jan;23(1):1-9. doi: 10.1016/j.soc.2013.09.001. Epub 2013 Nov 1. PMID 24267161
- [Background] Hong SM, Baek DH. A Review of Colonoscopy in Intestinal Diseases. Diagnostics (Basel). 2023 Mar 27;13(7):1262. doi: 10.3390/diagnostics13071262. PMID 37046479
- [Background] López Rosés L, Olivencia Palomar P. Colonoscopia. Rev Esp Enfermedades Dig. junio de 2008;100(6):372-372.
- [Background] Antoniou SA, Antoniou GA, Koutras C, Antoniou AI. Endoscopy and laparoscopy: a historical aspect of medical terminology. Surg Endosc. 2012 Dec;26(12):3650-4. doi: 10.1007/s00464-012-2389-y. Epub 2012 Jun 21. PMID 22717798
- [Background] Trujillo-Benavides O, Solana-Sentíes S, Aguilar-Mendoza J, Angulo-Molina D, Barrera-Torres H, Barreto-Zúñiga R, et al. Guía clínica de calidad en colonoscopia y polipectomía. Endoscopia. junio de 2021;33(2):54-74.
- [Background] Rivero-Sanchez L, Pellise M. [Bowel preparation for colonoscopy. Any significant progress on the horizon?]. Gastroenterol Hepatol. 2015 Apr;38(4):287-300. doi: 10.1016/j.gastrohep.2014.10.008. Epub 2014 Dec 10. Spanish. PMID 25499609
- [Background] Lorenzo-Zuniga V, Moreno-de-Vega V, Boix J. [Preparation for colonoscopy: types of scales and cleaning products]. Rev Esp Enferm Dig. 2012 Aug;104(8):426-31. doi: 10.4321/s1130-01082012000800006. Spanish. PMID 23039803
- See also: La alucinante evolución de la endoscopia — http://www.revistagastroenterologiamexico.org/es-pdf-X0375090601252936
- See also: Historia de la Endoscopia — https://www.amegendoscopia.org.mx/index.php/acerca/historia/145-historia-de-la-endoscopia